CLINICAL TRIAL: NCT03257462
Title: A Phase 2, Multiple-Dose, Dose-Escalation Study to Evaluate the Safety and Efficacy of SPR001 in Adults With Classic Congenital Adrenal Hyperplasia (CAH)
Brief Title: Study of SPR001 in Adults With Classic Congenital Adrenal Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spruce Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SPR001-201
Record Dates: First submitted 2017-08-15; First posted 2017-08-22 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Congenital Adrenal Hyperplasia; CAH - Congenital Adrenal Hyperplasia
Keywords: 17-hydroxyprogesterone
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A (Experimental): The first cohort of 9 patients will be administered SPR001 at dose strength of Dose A daily for 2 weeks, and escalating through Dose B per day for 2 weeks and Dose C per day for 2 weeks.
  Interventions: Drug: SPR001
- Cohort B (Experimental): Cohort B will begin enrollment after Cohort A has been fully enrolled. Starting dose selection and the stepwise dosing paradigm for Cohort B will be determined by an interim review of safety and PK/PD data from from Cohort A.
  Interventions: Drug: SPR001
- Cohort C (Experimental): Cohort C will begin enrollment after Cohort B has been fully enrolled. Starting dose selection and the stepwise dosing paradigm for Cohort C will be determined by an interim review of safety and PK/PD data from from Cohort A and B.
  Interventions: Drug: SPR001

INTERVENTIONS:
Drug: SPR001 — SPR001 Capsules

SUMMARY:
This is a multicenter Phase 2, multiple dose, dose escalation study to evaluate the safety, pharmacokinetics (PK), pharmacodynamics (PD), and efficacy of SPR001 in adult patients with classic congenital adrenal hyperplasia (CAH).

DETAILED DESCRIPTION:
This is a 6-week, multiple-dose, dose escalation study of SPR001 for the treatment of adults with classic CAH. After screening, eligible patients will be enrolled into a 6-week treatment period followed by a 4-week washout/safety follow-up period.

It is initially planned that up to approximately 18 patients in 2 dose cohorts will be enrolled. Additional patients or dose groups may be considered based upon specific safety, PK/PD, and/or efficacy findings, or if an active dose has not yet been reached.

SPR001 will be administered as an oral daily dose. Patients will undergo titration of SPR001 through three escalating dosage strengths at 2-week intervals. Patients will have overnight PK/PD assessments performed at baseline, which include an pre-dose overnight assessment and a post-dose overnight assessment for PK/PD following administration of the first dose. At the end of each 2-week dosing period, patients will return for single overnight visits for steady-state PK/PD assessments.

A follow-up outpatient visit will occur 30 days after their last dose.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18 or older.
* Documented diagnosis of classic CAH due to 21-hydroxylase deficiency
* Elevated 17-OHP at screening
* On a stable glucocorticoid replacement regimen for a minimum of 30 days

Exclusion Criteria:

* Clinically significant unstable medical condition, illness, or chronic disease
* Clinically significant psychiatric disorder.
* Clinically significant abnormal laboratory finding or assessment
* History of bilateral adrenalectomy or hypopituitarism
* Pregnant or nursing females
* Use of any other investigational drug within 30 days
* Unable to understand and comply with the study procedures, understand the risks, and/or unwilling to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2019-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spruce Chief Medical Officer, MD, Study Director — Spruce Biosciences; Richard Auchus, MD, PhD, Principal Investigator — University of Michigan
Locations (9):
- United States (9):
  - Spruce Biosciences Clinical Site, Orange, California
  - Spruce Biosciences Clinical Site, San Diego, California
  - Spruce Biosciences Clinical Site, Melbourne, Florida
  - Spruce Biosciences Clinical Site, Atlanta, Georgia
  - Spruce Biosciences Clinical Site, Indianapolis, Indiana
  - Spruce Biosciences Clinical Site, Ann Arbor, Michigan
  - Spruce Biosciences Clinical Site, Minneapolis, Minnesota
  - Spruce Biosciences Clinical Site, Las Vegas, Nevada
  - Spruce Biosciences Clinical Site, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sarafoglou K, Barnes CN, Huang M, Imel EA, Madu IJ, Merke DP, Moriarty D, Nakhle S, Newfield RS, Vogiatzi MG, Auchus RJ. Tildacerfont in Adults With Classic Congenital Adrenal Hyperplasia: Results from Two Phase 2 Studies. J Clin Endocrinol Metab. 2021 Oct 21;106(11):e4666-e4679. doi: 10.1210/clinem/dgab438. PMID 34146101
- See also: On-line clinical study-related information for patients, including pre-screening questionnaire. — http://cahclinicaltrial.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No participants enrolled in Period 4: Cohort D
Pre-assignment Details: A total of 24 subjects were enrolled into the study and 24 ICFs were signed. Two subjects were enrolled in more than one cohort: one subject was enrolled in both Cohorts A and C and one subject was enrolled in both in Cohorts A and B. Therefore, the total when adding Cohorts A+B+C = 26; however, 2 subject were the same, thus a total of 24 unique subjects participated and signed the ICFs.
Groups:
- Period 1: Cohort A: The first cohort of 9 patients underwent dose escalation through 3 dose levels of tildacerfont capsules, beginning with 200 mg QD for 2 weeks, then escalating to 600 mg QD/day for 2 weeks, then escalating to 1000 mg QD for 2 weeks with no washout between dose levels.
- Period 2: Cohort B: Cohort B will begin enrollment after Cohort A has been fully enrolled. Cohorts B, C, and D underwent a 2-week run-in period, a 2-week treatment period, and a 30-day washout and safety follow-up period. Cohort B was administered tildacerfont 200 mg BID during the treatment period.
- Period 3: Cohort C: Cohort C will begin enrollment after Cohort B has been fully enrolled. Cohorts B, C, and D underwent a 2-week run-in period, a 2-week treatment period, and a 30-day washout and safety follow-up period. Cohort C was administered tildacerfont 100 mg BID during the treatment period.
- Period 4: Cohort D: Cohort D will begin enrollment after Cohort C has been fully enrolled. Cohorts B, C, and D underwent a 2-week run-in period, a 2-week treatment period, and a 30-day washout and safety follow-up period. For Cohort D, the dose level and the frequency and timing of dosing were to be determined based on interim data from the previous cohorts, but the dose level of Cohort D was to be capped at 800 mg/day. Based on PK/PD results from Cohorts B and C, this cohort was not enrolled.
Period: Cohort A
Arm/Group | Period 1: Cohort A | Period 2: Cohort B | Period 3: Cohort C | Period 4: Cohort D
Started | 10 | 0 | 0 | 0
Completed | 9 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Period: Cohort B
Arm/Group | Period 1: Cohort A | Period 2: Cohort B | Period 3: Cohort C | Period 4: Cohort D
Started | 0 | 9 | 0 | 0
Completed | 0 | 8 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Discontinued due to Sponsor decision | 0 | 1 | 0 | 0
Period: Cohort C
Arm/Group | Period 1: Cohort A | Period 2: Cohort B | Period 3: Cohort C | Period 4: Cohort D
Started | 0 | 0 | 7 | 0
Completed | 0 | 0 | 6 | 0
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 24 unique subjects participated in the study; however, two subjects were enrolled in more than one cohort, one subject in Cohorts A and C and one subject in Cohorts A and B. For the subjects enrolled in more than 1 cohort, cohort totals/statistics reflect all baseline values.
Groups:
- Cohort A: The first cohort of 9 patients underwent dose escalation through 3 dose levels of tildacerfont capsules, beginning with 200 mg QD for 2 weeks, then escalating to 600 mg QD/day for 2 weeks, then escalating to 1000 mg QD for 2 weeks with no washout between dose levels.
- Cohort B: Cohort B will begin enrollment after Cohort A has been fully enrolled. Cohorts B, C, and D underwent a 2-week run-in period, a 2-week treatment period, and a 30-day washout and safety follow-up period. Cohort B was administered tildacerfont 200 mg BID during the treatment period.
- Cohort C: Cohort C will begin enrollment after Cohort B has been fully enrolled. Cohorts B, C, and D underwent a 2-week run-in period, a 2-week treatment period, and a 30-day washout and safety follow-up period. Cohort C was administered tildacerfont 100 mg BID during the treatment period.
- Cohort D: Cohort D will begin enrollment after Cohort C has been fully enrolled. Cohorts B, C, and D underwent a 2-week run-in period, a 2-week treatment period, and a 30-day washout and safety follow-up period. For Cohort D, the dose level and the frequency and timing of dosing were to be determined based on interim data from the previous cohorts, but the dose level of Cohort D was to be capped at 800 mg/day. Based on PK/PD results from Cohorts B and C, this cohort was not enrolled.
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D | Total
Number analyzed (Participants) | 10 | 8 | 6 | 0 | 24
Age, Categorical [Count of Participants; unit: Participants] — Population: Cohort A is reported separately from Cohorts B and C
  Participants
    Cohort A: number analyzed (Participants) | 10 | 0 | 0 | 0 | 10
    Cohort A: <=18 years | 0 | 0 | 0 | 0 | 0
    Cohort A: Between 18 and 65 years | 9 | 0 | 0 | 0 | 9
    Cohort A: >=65 years | 1 | 0 | 0 | 0 | 1
    Cohort B: number analyzed (Participants) | 0 | 8 | 0 | 0 | 8
    Cohort B: <=18 years | 0 | 0 | 0 | 0 | 0
    Cohort B: Between 18 and 65 years | 0 | 7 | 0 | 0 | 7
    Cohort B: >=65 years | 0 | 1 | 0 | 0 | 1
    Cohort C: number analyzed (Participants) | 0 | 0 | 6 | 0 | 6
    Cohort C: <=18 years | 0 | 0 | 0 | 0 | 0
    Cohort C: Between 18 and 65 years | 0 | 0 | 5 | 0 | 5
    Cohort C: >=65 years | 0 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Cohort A is reported separately from Cohorts B and C
  Participants
    Cohort A: number analyzed (Participants) | 10 | 0 | 0 | 0 | 10
    Cohort A: Female | 5 | 0 | 0 | 0 | 5
    Cohort A: Male | 5 | 0 | 0 | 0 | 5
    Cohort B: number analyzed (Participants) | 0 | 8 | 0 | 0 | 8
    Cohort B: Female | 0 | 1 | 0 | 0 | 1
    Cohort B: Male | 0 | 7 | 0 | 0 | 7
    Cohort C: number analyzed (Participants) | 0 | 0 | 6 | 0 | 6
    Cohort C: Female | 0 | 0 | 3 | 0 | 3
    Cohort C: Male | 0 | 0 | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Cohort A is reported separately from Cohorts B and C
  Participants
    Cohort A: number analyzed (Participants) | 10 | 0 | 0 | 0 | 10
    Cohort A: Hispanic or Latino | 3 | 0 | 0 | 0 | 3
    Cohort A: Not Hispanic or Latino | 7 | 0 | 0 | 0 | 7
    Cohort A: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
    Cohort B: number analyzed (Participants) | 0 | 8 | 0 | 0 | 8
    Cohort B: Hispanic or Latino | 0 | 2 | 0 |  | 2
    Cohort B: Not Hispanic or Latino | 0 | 6 | 0 |  | 6
    Cohort B: Unknown or Not Reported | 0 | 0 | 0 |  | 0
    Cohort C: number analyzed (Participants) | 0 | 0 | 6 | 0 | 6
    Cohort C: Hispanic or Latino | 0 | 0 | 1 |  | 1
    Cohort C: Not Hispanic or Latino | 0 | 0 | 5 |  | 5
    Cohort C: Unknown or Not Reported | 0 | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Cohort A is reported separately from Cohorts B and C
  Participants
    Cohort A: number analyzed (Participants) | 10 | 0 | 0 | 0 | 10
    Cohort A: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Cohort A: Asian | 0 | 0 | 0 | 0 | 0
    Cohort A: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Cohort A: Black or African American | 0 | 0 | 0 | 0 | 0
    Cohort A: White | 10 | 0 | 0 | 0 | 10
    Cohort A: More than one race | 0 | 0 | 0 | 0 | 0
    Cohort A: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
    Cohort B: number analyzed (Participants) | 0 | 8 | 0 | 0 | 8
    Cohort B: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Cohort B: Asian | 0 | 0 | 0 | 0 | 0
    Cohort B: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Cohort B: Black or African American | 0 | 0 | 0 | 0 | 0
    Cohort B: White | 0 | 8 | 0 | 0 | 8
    Cohort B: More than one race | 0 | 0 | 0 | 0 | 0
    Cohort B: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
    Cohort C: number analyzed (Participants) | 0 | 0 | 6 | 0 | 6
    Cohort C: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Cohort C: Asian | 0 | 0 | 0 | 0 | 0
    Cohort C: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Cohort C: Black or African American | 0 | 0 | 0 | 0 | 0
    Cohort C: White | 0 | 0 | 5 | 0 | 5
    Cohort C: More than one race | 0 | 0 | 1 | 0 | 1
    Cohort C: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 6 |  | 24
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (BMI) is a medical screening tool that measures the ratio of a subject's height to their weight to estimate the amount of body fat. BMI is calculated by using weight in kilograms (kg) divided by the square of height in meters (m2).
  kg/m^2 | 31.7 (11.80) | 30.4 (6.31) | 32.3 (5.67) |  | 31.4 (8.44)

OUTCOME MEASURES:

1. Primary Outcome: Safety of SPR001 in Patients With CAH
Description: Incidence of treatment-emergent adverse events, changes from Baseline to End-of-study in clinical laboratory parameters, physical examination findings, vital signs, ECG parameters
Time Frame: 6 weeks
Population: This full analysis set includes all subjects who received at least 1 dose of study drug. The FAS was used to analyze all safety data
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 10 | 9 | 7
Participants | 6 | 5 | 4

2. Primary Outcome: Change in 17-hydroxyprogesterone
Description: Change in 17-hydroxyprogesterone from Baseline to End-of-study. Results are expressed as mean percent change from baseline. Reductions in 17-OHP are indicators of better disease control.
Time Frame: Cohort A: Baseline/2a (Day -1-0), First dose/2b (Day 0-1), Visit 3 (Day 13-14), Visit 4 (Day 27-28), Visit 5 (Day 41-42). Cohort B and Cohort C: Visit 2 (Day 0-1), Visit 3 (Day 8), Visit 4 (Day 14-15), Visit 5 (Last dose +30d)
Population: Only subjects with both baseline and post baseline (week 2) assessments were summarized. Baseline values were collected at 8am on Visit 2a (Day -1) and post-baseline Week 2 values were collected at 8a on Visit 3, Visit 4, or Visit 5. A negative change indicates improvement.
Measure: Mean (Standard Deviation); unit: percentage of mean change from baseline
Groups:
- Cohort A - Dose A; Cohort A - Dose B; Cohort A - Dose C: The first cohort of 9 patients will be administered SPR001 at dose strength of Dose A daily for 2 weeks, and escalating through Dose B per day for 2 weeks and Dose C per day for 2 weeks.
  SPR001: SPR001 Capsules
Arm/Group | Cohort B | Cohort C | Cohort A - Dose A | Cohort A - Dose B | Cohort A - Dose C
Number analyzed (Participants) | 7 | 7 | 9 | 7 | 8
percentage of mean change from baseline | -47.79 (63.300) | -33.19 (41.604) | 22.16 (172.298) | -23.71 (64.146) | -13.79 (74.742)

3. Secondary Outcome: Changes in Pharmacodynamic (PD) Markers
Description: Changes in adrenocorticotropic hormone (ACTH) and androstenedione (A4) from Baseline to End-of-study are measured in patient serum. Results are expressed as a mean percentage change from baseline. A negative change indicates improvement.
Time Frame: Cohort A: Visit 2a (Day -1 to 0), Visit 2b (Days 0-1), Visit 3 (Day 13-14), Visit 4 (Day 27-28), Visit 5 (Day 41 to 42). Cohorts B+C: Visit 2 (Day 0-1), Visit 3 (Day 8), Visit 4 (Day 27-28), Visit 5 (+30 days after last dose)
Population: Only subjects with both baseline and post baseline (week 2) assessments were summarized. Baseline values were collected at 8am on Visit 2a (Day -1) and post-baseline Week 2 values were collected at 8a on Visit 3, Visit 4, or Visit 5.
Measure: Mean (Standard Error); unit: percentage of mean change from baseline
Groups:
- PD Population Cohort B: Cohort B will begin enrollment after Cohort A has been fully enrolled. Starting dose selection and the stepwise dosing paradigm for Cohort B will be determined by an interim review of safety and PK/PD data from from Cohort A.
  SPR001: SPR001 Capsules
- PD Population Cohort C: Cohort C will begin enrollment after Cohort B has been fully enrolled. Starting dose selection and the stepwise dosing paradigm for Cohort C will be determined by an interim review of safety and PK/PD data from from Cohort A and B.
  SPR001: SPR001 Capsules
- PD Population - Cohort A Dose A; PD Population Cohort A - Dose B; PD Population - Cohort A - Dose C: The first cohort of 9 patients will be administered SPR001 at dose strength of Dose A daily for 2 weeks, and escalating through Dose B per day for 2 weeks and Dose C per day for 2 weeks.
  SPR001: SPR001 Capsules
Arm/Group | PD Population Cohort B | PD Population Cohort C | PD Population - Cohort A Dose A | PD Population Cohort A - Dose B | PD Population - Cohort A - Dose C
Number analyzed (Participants) | 8 | 7 | 10 | 9 | 9
percentage of mean change from baseline
  Adrenocorticotropic hormone (ACTH) | -26.05 (54.807) | 16.66 (120.211) | -28.53 (53.834) | -67.60 (32.100) | -36.83 (48.510)
  Androstenedione (A4) | -1.58 (101.458) | -30.17 (35.055) | -12.12 (47.381) | -33.18 (36.465) | -28.93 (45.167)

4. Secondary Outcome: Pharmacokinetic Parameter - Maximum Plasma Concentration (Cmax)
Description: To evaluate the pharmacokinetic (PK) parameter of maximum plasma concentration (Cmax) of SPR001 in patients with CAH.
Time Frame: Serial PK sampling was performed at the end of the 2 weeks for all cohorts and dose levels
Measure: Mean (Standard Deviation); unit: ng/dL
Groups:
- PK Population Cohort B: Cohort B will begin enrollment after Cohort A has been fully enrolled. Starting dose selection and the stepwise dosing paradigm for Cohort B will be determined by an interim review of safety and PK/PD data from from Cohort A.
  SPR001: SPR001 Capsules
- PK Population Cohort C: Cohort C will begin enrollment after Cohort B has been fully enrolled. Starting dose selection and the stepwise dosing paradigm for Cohort C will be determined by an interim review of safety and PK/PD data from from Cohort A and B.
  SPR001: SPR001 Capsules
- PK Population - Cohort A Dose A; PK Population Cohort A - Dose B; PK Population - Cohort A - Dose C; PK Population Cohort A - Dose A (After single dose): The first cohort of 9 patients will be administered SPR001 at dose strength of Dose A daily for 2 weeks, and escalating through Dose B per day for 2 weeks and Dose C per day for 2 weeks.
  SPR001: SPR001 Capsules
Arm/Group | PK Population Cohort B | PK Population Cohort C | PK Population - Cohort A Dose A | PK Population Cohort A - Dose B | PK Population - Cohort A - Dose C | PK Population Cohort A - Dose A (After single dose)
Number analyzed (Participants) | 8 | 7 | 10 | 10 | 9 | 10
ng/dL | 411.25 (130.107) | 200.96 (132.262) | 283.69 (150.116) | 719.30 (325.056) | 892.56 (289.272) | 96.35 (86.1)

5. Secondary Outcome: Pharmacokinetic Parameter - Area Under the Concentration-time Curve (AUC)
Description: To evaluate the PK parameter of area under the concentration-time curve (AUC) of SPR001 in patients with CAH
Time Frame: For Cohort A, serial blood collections were made for PK measurements on Day 1 for 200 mg SD and at Week 2 for all QD dose levels. In Cohorts B and C, serial blood samples were drawn for PK measurements at the end of the 2-week treatment period.
Measure: Mean (Standard Deviation); unit: ng*hr/dL
Groups:
- PK Population Cohort B: 200 mg BID capsules
- PK Population Cohort C: 100 mg BID capsules
- PK Population - Cohort A Dose A: 200 mg QD capsules
- PK Population Cohort A - Dose B: 600 mg QD capsules
- PK Population - Cohort A - Dose C: 1000 mg QD capsules
- PK Population Cohort A - Dose A (After single dose): 200 mg SD capsules
Arm/Group | PK Population Cohort B | PK Population Cohort C | PK Population - Cohort A Dose A | PK Population Cohort A - Dose B | PK Population - Cohort A - Dose C | PK Population Cohort A - Dose A (After single dose)
Number analyzed (Participants) | 8 | 7 | 10 | 10 | 9 | 10
ng*hr/dL | 2975.968 (970.6) | 1425.582 (941.9188) | 1474.162 (642.6) | 4449.263 (1826.4801) | 6212.983 (2051.9077) | 421.539 (331.54)

ADVERSE EVENTS:
Time Frame: 6-week treatment period followed by a 4-week washout/safety follow-up period
Groups:
- Cohort A - Dose A: The first cohort of 9 patients will be administered SPR001 at dose strength of Dose A daily for 2 weeks and escalating through Dose B per day for 2 weeks and Dose C per day for 2 weeks.
  SPR001: SPR001 Capsules
- Cohort A - Dose B; Cohort A - Dose C: The first cohort of 9 patients will be administered SPR001 at dose strength of Dose A daily for 2 weeks and escalating through Dose B per day for 2 weeks and Dose C per day for 2 weeks.
- Cohort B: Cohort B will begin enrollment after Cohort A has been fully enrolled. Starting dose selection and the stepwise dosing paradigm for Cohort B will be determined by an interim review of safety and PK/PD data from from Cohort A. One subject from Cohort A was allowed to enroll in Cohort B.
  SPR001: SPR001 Capsules
- Cohort C: Cohort C will begin enrollment after Cohort B has been fully enrolled. Starting dose selection and the stepwise dosing paradigm for Cohort C will be determined by an interim review of safety and PK/PD data from from Cohort B. One subject from Cohort A was allowed to enroll in Cohort C.
  SPR001: SPR001 Capsules
Arm/Group | Cohort A - Dose A | Cohort A - Dose B | Cohort A - Dose C | Cohort B | Cohort C
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/9 | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 6/10 | 3/10 | 3/9 | 5/9 | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - Dose A (N=10) | Cohort A - Dose B (N=10) | Cohort A - Dose C (N=9) | Cohort B (N=9) | Cohort C (N=7)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hunger (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Salivary gland enlargement (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT03257462/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT03257462/SAP_001.pdf